CLINICAL TRIAL: NCT06981897
Title: Impact Of Early Cognitive Rehabilitation On Functional Outcomes Following Moderate Traumatic Brain Injury
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Amany Saadallah Hassan Mobarez (Other)
Responsible Party: Sponsor-Investigator, Amany Saadallah Hassan Mobarez, Senior physiotherapist, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TBI
Record Dates: First submitted 2025-05-03; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: TBI (Traumatic Brain Injury)
Keywords: COGNITION / TBI/
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Patient Positioning; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Seventeen Patients in study group will receive selected physical therapy program (Chest care exercise, passive movement of the four limbs) in addition to early cognitive therapy program
  Interventions: Behavioral: early cognitive therapy program in addition to selected physical therapy program (positioning, chest care exercise).; Behavioral: selected physical therapy program (Chest care exercise, passive movement of the four limbs) in addition to early cognitive therapy program; Behavioral: Control group
- Control group (Experimental): Seventeen Patients in control group will receive selected physiotherapy program only Chest care exercise, passive movement of the four limbs.
  Interventions: Behavioral: selected physical therapy program (Chest care exercise, passive movement of the four limbs) in addition to early cognitive therapy program; Behavioral: Control group

INTERVENTIONS:
Behavioral: early cognitive therapy program in addition to selected physical therapy program (positioning, chest care exercise). — A.Positioning for head injury patients
  B.Chest clearance intervention
  C.Procedure for cognitive therapy All these exercises are given to patients even when they are on ventilator support of around 20-30 minutes six days /week .
  1. coma stimulation incorporated with cognition training such as : i. Multimodal Sensory stimulation, including :
     1. Visual
     2. Auditory
     3. Olfactory
     4. Gustatory
     5. Tactile- Administered by rubbing different textures like satin, silk, fur, smooth metal, sandpaper, or cool or warm items over the patient's body surfaces.
     ii. Calling out their names, using patient's relatives help for transferring were used for improving the cognition and conscious levels.
  2. Kinesthetic Stimulation
     1. Passive movements
     2. Joint approximation Each movement two times, allowing 1 minute to respond. This will be performed either in bed or in the wheelchair, one extremity at a time.
  Arms: study group
Behavioral: selected physical therapy program (Chest care exercise, passive movement of the four limbs) in addition to early cognitive therapy program — The patient was placed in a comfortable position with a head-up position Passive range of movement for all four limbs & positioning for head injury patients,. Joint approximation and Chest clearance intervention and Procedure for cognitive therapy
  Multimodal Sensory stimulation, including :
  Visual Auditory- Olfactory-. Gustatory- Tactile- Calling out their names, using patients relative help for transferring were used for improving the cognition and conscious levels.
Behavioral: Control group — The patient was placed in a comfortable position with a head-up position , Passive range of movement for all four limbs and positioning for head injury patients,. Joint approximation and Chest clearance intervention

SUMMARY:
Purpose of the study:

This study aims to detect the impact of early cognitive rehabilitation on functional outcomes with patients following moderate traumatic brain injury.

DETAILED DESCRIPTION:
Intensive care unit (ICU) hospitalization saves lives but often costs ICU survivors, who often experience cognitive impairment and physical and functional disabilities. Early physical rehabilitation improves chances of regaining pre-hospital functional status, but early cognitive rehabilitation for these patients remains unexplored Traumatic brain injury occurs from violent blows or objects, causing physical and psychological effects. Signs may appear immediately or days later, affecting the brain's function and functioning . Traumatic Brain Injury (TBI) impacts health and quality of life, with unpredictable prognosis. Exercise is crucial for neuroplasticity and brain rewiring.The Glasgow Coma Scale, published in 1974, measures impaired consciousness in acute medical and trauma patients using eye-opening, motor, and verbal responses. It provides a clear, communicable picture of a patient's state.

The Rancho Los Amigos Scale (RLAS) is a medical assessment tool for individuals recovering from closed head injuries, including traumatic brain injuries. It evaluates cognitive and behavioral presentations as they emerge from coma, comparing patients' state of consciousness and reliance on assistance .

The Functional Independence Measure (FIM) is an 18-item assessment tool for evaluating patients' functional status in rehabilitation after stroke, traumatic brain injury, spinal cord injury, or cancer. It evaluates self-care, continence, mobility, transfers, communication, and cognition, with each item rated 1-7 .

ELIGIBILITY:
Inclusion Criteria:

1. Both Genders.
2. Moderate traumatic brain injury patients will be included with GCS score 9-12.
3. Patients' age 18 years old and more .
4. All patients must be medically stable post trauma.

Exclusion Criteria:

1. children under 18 years old .
2. Previous cerebral infarction and intracranial space-occupying lesions.
3. Patients with cancer and major underlying illnesses.
4. Patients with diffuse axonal damage.
5. Incomplete clinical and imaging data
6. Patient with other neurological deficits or orthopedic abnormalities that causing disability.
7. Patients with serious psychiatric pathology or mentally. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Glassgow Coma Scale | evaluation post every week at first two weeks of treatment at ICU after injury
  being aware of and responsive to one's surroundings a person's awareness or perception of something wchich evaluated by glassgow coma scale .No eye opening / 1 No eye opening Eye opening to pain / 2 Eye opening to pain Eye opening to sound / 3 Eye opening to sound Eyes open spontaneously / 4 Eyes open spontaneously Best verbal response
  None / 1 None Moans in response to pain / 2 Incomprehensible sounds Cries in response to pain / 3 Incomprehensible words Irritable/cries / 4 Confused Coos and babbles / 5 Orientated - appropriate Best motor response
  No motor response / 1 No motor response. Abnormal extension to pain / 2 Abnormal extension to pain Abnormal flexion to pain / 3 Abnormal flexion to pain Withdrawal to pain / 4 Withdrawal to pain Withdraws to touch / 5 Localises to pain Moves spontaneously and purposefully / 6 Obeys commands
Rancho Los amigos scale | evaluation post every week at first two weeks of treatment at ICU after injury
  evauating of conscious intellectual activity such as thinking, reasoning or remembering wchich evaluated by The Rancho Los Amigos Scale (RLAS), Level I No response/total assistance Level II Generalised response/total assistance Level III Localised response/total assistance Level IV Confused and agitated/max assist Level V Confused, inappropriate non-agitated/max assist Level VI Confused, appropriate/ mod assist Level VII Automatic, appropriate/ min assist for ADLs Level VIII Purposeful, appropriate/ stand by assist Level IX Purposeful, appropriate/ stand by assist on request Level X Purposeful, appropriate/ modified independent
Functional Independence Measure | evaluation post every week at first two weeks of treatment at ICU after injury
  assess and grade the functional status of a person based on the level of assistance he or she requires wchich evaluated by functional Independence Measure (FIM)scored on a 7-point Likert scale, and the score indicates the amount of assistance required to perform each item (1 = total assistance in all areas, 7 = total independence in all areas). The ratings are based on performance rather than capacity and can be acquired by observation, patient interview, telephone interview or medical records. The developers of the FIM recommend that the scoring be derived by consensus with a multi-disciplinary team.

CONTACTS AND LOCATIONS:
Overall Officials: Eman S. M. Fayez, Prof., Study Director — Professor of Physical Therapy , Cairo University; Ahmad A.S. El-Fiki, Prof., Study Director — Professor of Neurosurgery , Cairo University; Maged A. Gomaa, Ass.Prof., Study Director — Associate professor of psychiatry, Cairo University
Locations (3):
- Egypt (3):
  - Cairo University hospital, Cairo, Manial
  - Kasr Al-Ainy Emergency Hospital185, Cairo
  - Cairo University hospital, Cairo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: a systematic review following the PRISMA protocol primarily to identify publications that assessed any links between mechanical ventilation (MV) and either cognitive impairment or brain insult, independent of underlying medical conditions. — https://www.biomedcentral.com/

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT06981897/Prot_SAP_ICF_000.pdf